CLINICAL TRIAL: NCT00746304
Title: Long-Term Outcomes in the Treatment of Infantile and Acquired Esotropia With Botulinum Toxin
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Tsai Tzu-Hsun, National Taiwan University Hospital
Other Study IDs: 200709002R
Record Dates: First submitted 2008-08-31; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2007-09

CONDITIONS: Esotropia
Keywords: botulinum; esotropia
MeSH Terms: conditions — Esotropia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: infantile esotropia
- 2: acquired esotropia

SUMMARY:
To investigate long-term treatment outcomes of patients receiving botulinum toxin A therapy for infantile and acquired esotropia.

DETAILED DESCRIPTION:
Participants: 164 patients with infantile esotropia and 89 patients with acquired esotropia.

Methods: Patients were injected with botulinum toxin into two medial rectus muscles and followed from 1992 to 2005. Patients were evaluated at 1 week, 2, 6 and 12 months, and then yearly post-injection.

Main Outcome Measures: Degree of motor alignment, recurrence rate, incidence of stereopsis, and dissociated vertical deviation along with complications.

ELIGIBILITY:
Inclusion Criteria:

* infantile esotropia and acquired esotropia

Exclusion Criteria:

* exotropia, high AC/A ratio accommodative esotropia, patients with neurological deficit including cerebral palsy, Down syndrome and mental retardation, and ocular anomalies including retinopathy of prematurity. Patients lost to follow-up at 6 months or less after the last injection were also excluded.

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 373 patients with strabismus were treated with botulinum toxin injection by a single surgeon (AH Wang) at the Department of Ophthalmology, National Taiwan University Hospital, Taipei, Taiwan from 1992 to 2005.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Degree of motor alignment, recurrence rate, incidence of stereopsis, and dissociated vertical deviation along with complications. | Before treatment, weekly after the treatment, and monthly after motor alignment

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Hsun Tsai, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan